CLINICAL TRIAL: NCT07022951
Title: The Million Anesthesia Cases Study (MACS) - Retrospective and Prospective Characterization of Perioperative Fasting Practices and Their Effects on Clinical Outcomes
Brief Title: The Million Anesthesia Cases Study (MACS) - a Cohort Study of Preoperative Fasting and Perioperative Outcomes
Acronym: MACS
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Alexander Nagrebetsky, MD MSc, Physician-Investigator, Massachusetts General Hospital
Other Study IDs: 2023P001743
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Anesthesia; Sedation; Monitored Anesthesia Care; Procedure; Surgery, Day; Surgery; Surgery Scheduled; Fasting Before Operation; Aspiration; Gastric Contents, Anesthesia
Keywords: preoperative fasting; perioperative pulmonary aspiration; perioperative complications; postoperative nausea and vomiting; perioperative hypoglycemia; perioperative hyperglycemia; perioperative hypotension; myocardial injury after noncardiac surgery; perioperative acute kidney injury; clear liquid fasting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who receive anesthesia care
  Interventions: Other: Preoperative fasting

INTERVENTIONS:
Other: Preoperative fasting — This cohort study assesses the duration of preoperative fasting and its clinical effects

SUMMARY:
Perioperative fasting has historically been viewed as a low-risk intervention. However, preliminary data indicate that perioperative loss of nutrition and fluids is likely harmful. This study intends to characterize perioperative fasting practices and their potential effects on clinical outcomes through possible effects on patient well-being (anxiety, hunger, thirst), physiology (hypovolemia, hypotension), perioperative aspiration, etc. We hypothesized that in addition to known adverse effects on patients' well-being, prolonged preoperative fasting adversely affects circulating blood volume-related (hypotension, decreased urine output etc.) and glucose metabolism-related (e.g., hypo/hyperglycemia) perioperative physiology.

Additional knowledge on the potential adverse effects of preoperative fasting will inform preoperative fasting policies and research interventions that are relevant to hundreds of millions of patients subjected to preoperative/preprocedural fasting worldwide each year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic or therapeutic procedure with anesthesia care (general anesthesia, regional anesthesia, sedation, or a combination of the above)

Exclusion Criteria:

* Not receiving anesthesia care
* Lack of medical record data in Epic electronic medical record system

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will include all anesthesia cases at participating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 1200000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of fasting-related perioperative complications: pulmonary aspiration; patient well-being (anxiety, hunger, thirst); circulating blood volume-related complications (hypotension, myocardial and kidney injury); dysglycemia. | Perioperative period - while patient is located in the preoperative area, procedure area, or recovery area.

CONTACTS AND LOCATIONS:
Locations (1):
- Mass General Brigham, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No